CLINICAL TRIAL: NCT06122675
Title: Cerebellar Deep Brain Stimulation for Severe Combined Movement Disorders and Spasticity in Children and Young Adults with Cerebral Palsy
Brief Title: Cerebellar Deep Brain Stimulation for Movement Disorders in Cerebral Palsy in Children and Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Marta San Luciano Palenzuela, MD, Associate Professor, Neurology, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-37182; UH3NS128297-01A1 (NIH)
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-02

CONDITIONS: Dyskinetic Cerebral Palsy; Dystonic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The differences in primary outcome scores are calculated while on intervention (effective stimulation) versus placebo (sham stimulation), using an N-of-1 trial design. Each N-of-1 trial consists of a baseline assessment prior to DBS surgery (4 weeks), DBS surgery and open label phase to determine optimal stimulation settings (20 weeks), followed by a randomized three-cycle sequence of paired 8-week exposure periods, with each pair including intervention then placebo or vice versa (24 weeks). The DBS intervention exposure will be at the personalized optimal stimulation settings determined during the open-label phase.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Effective stimulation (Active Comparator): All participants will receive deep brain stimulation (DBS) in the cerebellum. For the first 20 weeks, every participant undergoes an open label phase to titrate stimulation and determine optimal stimulation settings. Following that phase, each participant starts three cycles of randomized, paired 8-week exposure periods, each pair including effective stimulation followed by sham stimulation, or vice versa. Effective stimulation will be the optimal stimulation settings determined during the open label phase.
  Interventions: Device: DBS
- Sham stimulation (Sham Comparator): Sham stimulation will be settings at low amplitude (0.1mA) known to be ineffective.
  Interventions: Device: DBS

INTERVENTIONS:
Device: DBS — Implanted in the cerebellum.
  Other Names: Medtronic Percept

SUMMARY:
The purpose of this study is to test the safety of placing Deep Brain Stimulators (DBS) in a part of the brain called the cerebellum and using electrical stimulation of that part of the brain to treat movement symptoms related to cerebral palsy. Ten children and young adults with dyskinetic cerebral palsy will be implanted with a Medtronic Percept Primary Cell Neurostimulator. We will pilot videotaped automated movement recognition techniques and formal gait analysis, as well as collect and characterize each subject's physiological and neuroimaging markers that may predict hyperkinetic pathological states and their response to therapeutic DBS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DCP (dystonic and/or choreoathetotic cerebral palsy) with or without comorbid spasticity, with a clear history of hypoxic ischemic brain injury preceding motor symptoms made by a pediatric neurologist, with supporting MRI findings.
* Age 7-25 at the time of surgery.
* Gross Motor Function Classification System (GMFCS) Levels II-V.
* History of appropriate therapy with oral medications with inadequate relief as determined by a movement disorders or pediatric neurologist. Prior history of selective dorsal rhizotomy is allowed.
* Patient and family have requested surgical intervention with DBS for their movement disorder.
* No gross cerebellar abnormalities observed and reported on structural MRI.
* Written informed consent and written/verbal assent for those younger than 18 years of age.
* Ability to comply with study follow-up visits for brain recordings, neuroimaging and testing of sham and effective stimulation and clinical assessments.

Exclusion Criteria:

* Coagulopathy, uncontrolled epilepsy, severe cardiopulmonary or gastrointestinal conditions, or other medical conditions considered to place the patient at elevated risk for surgical complications.
* Pregnancy: all women of child-bearing potential will be required to have a negative urine pregnancy test prior to undergoing their surgical procedure.
* Exclusion of genetic mimics of cerebral palsy: exclusion of conditions that manifest with a clinical syndrome similar to CP, in the absence of documented risk factors or neuroimaging findings consistent with a history of brain injury or congenital cerebral malformation. Work up may include comparative genomic hybridization (CGH) microarray and multi-gene panel and/or whole genome or whole exome sequencing.)
* Severe fixed contractions and skeletal deformities that would preclude determination of improvement.
* Traumatic brain injury (i.e., non-accidental trauma) or history of infectious or autoimmune encephalitis.
* Requirement of diathermy, electroconvulsive therapy or transcranial magnetic stimulation.

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Average total (global index) Movement Disorder-Childhood Rating Scale 4-18 Revised (MD-CRS 4-18-R) scores | Evaluated weekly during randomized blinded phase (total of 3 months in each condition, sham stimulation and effective stimulation).
  This is the primary motor outcome measure. It is the Movement Disorder-Childhood Rating Scale 4-18 Revised (MD-CRS 4-18 R). The MD-CRS 4-18 R is a validated tool aimed to evaluate movement disorders in developmental age. It is particularly useful for rating the severity of movement disorders in dyskinetic cerebral palsy. It scored based on two parts. Part I: General Assessment has a minimum total score of 0 (no impairment) and a maximum total score of 60 (maximal impairment). Part II: MD Assessment has a minimum total score of 0 (movement disorder is absent) and a maximum total score of 28 (maximal movement disorder presence).
Average total standardized Caregiver Priorities & Child Health Index of Life with Disabilities (CPCHILD) scores | Evaluated weekly during randomized blinded phase (total of 3 months in each condition, sham stimulation and effective stimulation).
  This is the primary Quality of Life (QOL) outcome measure. It is the Caregiver Priorities & Child Health Index of Life with Disabilities (CPCHILD) scale. The CPCHILD is a reliable and valid measure of caregivers' perspectives on health status, functional limitations, and well-being of patients with severe CP, including those individuals who are non-verbal and non-ambulatory. Because many children suffering with CP are severely affected in many areas of their lives including activities of daily living, communication, mobility and overall health, there is an imperative to evaluate new interventions, especially invasive and resource-intensive ones such as DBS, using outcomes that are more meaningful to patients and their caregivers. Scores for each domain and for the total survey are standardized and range from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Marta San Luciano Palenzuela, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] San Luciano M, Oehrn CR, Wang SS, Tolmie JS, Wiltshire A, Graff RE, Zhu J, Starr PA. Protocol for combined N-of-1 trials to assess cerebellar neurostimulation for movement disorders in children and young adults with dyskinetic cerebral palsy. BMC Neurol. 2024 Apr 29;24(1):145. doi: 10.1186/s12883-024-03633-z. PMID 38684956
- [Derived] San Luciano M, Oehrn CR, Wang SS, Tolmie JS, Wiltshire A, Graff RE, Zhu J, Starr PA. Protocol for combined N-of-1 trials to assess cerebellar neurostimulation for movement disorders in children and young adults with dyskinetic cerebral palsy. Res Sq [Preprint]. 2024 Apr 1:rs.3.rs-4077387. doi: 10.21203/rs.3.rs-4077387/v1. PMID 38645256